CLINICAL TRIAL: NCT03259724
Title: The Effect of Non-Viscous Fibre Supplementation on Glycemic Control in Individuals With Diabetes Mellitus: A Systematic Review & Meta-analysis of RCTs
Brief Title: The Effect of NVFS on GC in Individuals With DM: SR & MA of RCTs
Acronym: NVFS&GC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: NVFS&GC Meta
Record Dates: First submitted 2017-08-21; First posted 2017-08-24 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Purpose of Study (The Effect of Non-Viscous Fibre Supplementation on Glycemic Control (NVFS & GC) in Individuals with Diabetes Mellitus.

Regardless of the remarkable advancement in pharmacotherapy, diabetes mellitus remains a major concern with more than 300 millions living with its complications including CVD. Nutrition is a cornerstone in diabetes management, and increasing total dietary fibre have been shown to decrease HbA1c, fasting glucose, fasting insulin, fructosamine, and HOMA-IR. However, the main underlying mechanism is still not fully understood, and the specific type and proportion of fibre supplementation to be recommended for such individuals is still controversial.

Currently, the available findings/ results from small RCTs are inconsistent. The systematic review method depends on combining data from many small studies in order a pooled estimate of the pooled effect. The purpose of this study is to conduct a systematic review and meta-analysis of randomized controlled trials (RCTs) assessing the effect of non-viscous fibre supplementation on fasting glucose and insulin in individuals with diabetes mellitus. We hope the findings of this study will play a role in developing the nutritional guidelines for individuals with diabetes mellitus.

DETAILED DESCRIPTION:
Background: High fibre diets have been recommended for individuals with diabetes mellitus. However, the findings on the effect of non-viscous fibre supplementation such as inulin, wheat bran and resistant starch on glycemic control in individuals with diabetes are inconsistent.

Objective: In order to improve the evidence-based guidelines for diabetes mellitus, we will conduct a systematic review and meta-analysis to assess evidence from randomized controlled trials (RCTs) on the effect of non-viscous fibre supplementation on glycemic control in individuals with diabetes.

Design: Cochrane handbook for systematic review of interventions will be used for planning and conducting this meta-analysis. The reporting will follow the Preferred Reporting Items for Systematic Reviews and Meta-analysis (PRISMA) guidelines.

Data sources: MEDLINE, EMBASE, the Cochrane Central Register for Controlled Trials will be searched using appropriate pre-determined search terms.

Study selection: All the included trials must be randomized, controlled, with duration of ≥ 3 weeks investigating the effect of supplementing diet with non-viscous fiber on glycemic control outcomes in individuals with diabetes mellitus. Acute studies, non-randomized, not appropriately controlled studies will be excluded. Both isocaloric and non-isocaloric will be included.

Data extraction: Two independent reviewers will extract information about fiber type, sample size, subject characteristics, dose, follow-up, composition of the background diets, and statistical analyses. Mean±SEM values will be extracted for all outcomes. Standard computation and imputation will be used to derive all missing variance data. Risk of bias and study quality will be assessed using the Cochrane Risk of Bias Tool and the Grading of Recommendations Assessment, Development and Evaluation (GRADE), respectively.

Outcome: This meta-analysis will assess a set of outcomes related to glycemic control in individuals with diabetes mellitus. These outcomes are: (1) glycated hemoglobin A1c (HbA1c) or (2) fructosamine, (3) fasting glucose (FG), (4) fasting insulin (FI), and (5) Homeostasis model assessment of insulin resistance (HOMA-IR).

Data synthesis: Pooled analysis will be conducted using the Generic Inverse Variance method. Rand-effects models will be used even in the absence of statistical significant between-study heterogeneity because they yield more conservative summary effect estimates in the presence of residual heterogeneity. Heterogeneity will be assessed using Cochran's Q test and quantified by the I2 statistic. Sensitivity and subgroup analyses will be used to explore sources of heterogeneity. A priori subgroup analyses include study design, does, fiber type, follow-up (duration), baseline values, study quality, food matrix, and composition of the background diet. The significance of subgroup analyses will be assessed using meta-regression analyses. Publication bias will be assessed using the inspection of funnel plots and application of Egger's and Begg's tests.

Knowledge translation plan: Results will be shared through traditional, national, and international scientific meetings and they may be submitted to high impact factor journals for publication.

Significance: We hope the results of this study will play a role in improving the guidelines/ recommendations for individuals with diabetes mellitus by raising the awareness towards viscous fiber consumption among health providers, patients, and industry. Hopefully, this study will aid in guiding future research in the dietary fiber field.

ELIGIBILITY:
Inclusion Criteria:

* Randomized
* Properly controlled
* ≥ 3 weeks
* Non-viscous fibre supplementation intervention
* Glycemic control endpoints
* Individuals with DM

Exclusion Criteria:

* Non-randomized
* Not controlled
* < 3 weeks
* Viscous fibre supplementation as intervention or placebo
* Healthy individuals or individuals with conditions other than DM

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with T1DM or T2DM
Sampling Method: Probability Sample
Enrollment: 514 (Estimated)
Dates: Start 2017-01-30 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-08-30 (Estimated)

PRIMARY OUTCOMES:
HbA1c | ≥ 3 weeks
  Glycated Hemoglobin A1C

SECONDARY OUTCOMES:
FG | ≥ 3 weeks
  Fasting Glucose
FI | ≥ 3 weeks
  Fasting Insulin
Fructomsamine | ≥ 3 weeks
HOMA-IR | ≥ 3 weeks
  Insulin Resistance

CONTACTS AND LOCATIONS:
Locations (1):
- The Toronto 3D Knowledge Synthesis and Clinical Trials Unit, Clinical Nutrition and Risk Factor Modification Centre, Toronto, Ontario, Canada